CLINICAL TRIAL: NCT06168266
Title: Effects of Smart Eccentric Exercise Training on Lymphocyte Immunity and Erythrocyte Rheology in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Eccentric Exercise Training in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH111246
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: COPD
Keywords: COPD; Eccentric Exercise Training; Lymphocytes; Mitochondria; Erythrocytes; Rheology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Undergoing conventional treatment
  Interventions: Other: conventional group
- Intervention Group: eccentric cycling exercise (Experimental): Received eccentric cycling exercise
  Interventions: Device: Eccentric bike

INTERVENTIONS:
Device: Eccentric bike — Received eccentric cycling exercise
  Arms: Intervention Group: eccentric cycling exercise
Other: conventional group — Received conventional treatment
  Arms: Control group

SUMMARY:
The goal of this study is to design eccentric exercise strategies for COPD patients to comprehensively improve their cardiopulmonary/muscular fitness, immune and hemorheological functions, and quality of life, thereby improving the prognosis of their disease.

DETAILED DESCRIPTION:
Background： The pathological process of COPD is often accompanied by a decrease in the number and distribution of immune cells in the blood, resulting in immune dysfunction, persistent, multiple infections, and systemic inflammation. Furthermore, the high oxidative stress induced by COPD may also depress the rheological properties of erythrocytes and cause secondary circulatory dysfunction. However, ventilatory limitation and decreased muscle function in COPD patients limit the patients to perform higher-effort exercise therapy. Compared with concentric exercise, eccentric exercise can effectively improve health-related physical fitness and quality of life under lower cardiorespiratory and metabolic loads.

Study Design： This is a three-year project in single center; COPD patients with GOLD grades are recruited in the first year, and then divided into four groups according to GOLD severity grades, and 50 subjects are expected to be recruited; In the second and third year, 120 COPD patients with GOLD grades were recruited.

Methods： This study is expected to recruit 170 subjects, and it will be conducted in the pulmonary rehabilitation treatment room. In the first year, 50 COPD patients with GOLD grade will be recruited, and 20 mL of the venous blood will be drawn during rest for follow-up blood analysis. After that, each subject will perform a serious of functional test, including Six-minute walk test, Timed up-and-go test, Stairs ascending and descending walking time, cardiopulmonary exercise test and isokinetic muscle test. In the second and third year, 60 COPD patients will be recruited respectively, and they will be randomly assigned to the eccentric exercise training and control groups (general care group), each group will carry out the experiment including three stages: control period, training period (and general care group) and maintenance period. During the training period, the eccentric exercise training group will perform 36 eccentric cycling exercises with progressive exercise intensity for 12 weeks, each session about 40 minutes (including 5-min warm-up, 30-min exercise and 5-min relaxation). In the control period, maintenance period and general care group, no exercise intervention will be performed; and in these three experimental periods, 4 functional tests and 4 resting blood draws will be performed.

Effect： This project expects that after 12 weeks of intelligent eccentric exercise training, COPD patients will effectively improve their health-related fitness and quality of life under lower cardiorespiratory and metabolic loads, and will benefit from peripheral blood lymphocytes. Changes in lymphocyte immunity and erythrocyte rheology, to classfy the biological indicators of the course of COPD.

Key words： COPD, Eccentric Exercise Training, Lymphocytes, Mitochondria, Erythrocytes, Rheology

ELIGIBILITY:
Inclusion Criteria:

* Having undergone pulmonary rehabilitation for more than 3 months
* Sign the written informed consent form
* FEV1/FVC < 0.70
* Approval for exercise training granted by a specialist physician's assessment
* Specialist physician's approval for exercise training

Exclusion Criteria:

* Existing of tracheostomy
* Those who use oxygen therapy or ventilator at home
* Severe heart failure (NYHA III-IV)
* Neuromuscular disease
* Acute exacerbation within the past three months
* Those who are unable to cooperate with the cardiopulmonary exercise test
* Taking anticoagulant medications
* Other conditions restricting exercise for over a year
* Recent or planned significant cardiovascular surgery or intervention
* Current or planned pregnancy within the next year
* Planned heart transplant within the next six months
* Heart failure due to uncorrectable valvular heart disease, congenital heart disease or obstructive cardiomyopathy
* Inadequate ICD settings for exercise heart rate
* Other exercise contraindications: unstable angina, uncontrolled blood pressure, orthostatic hypotension with symptoms, severe aortic stenosis, acute discomfort or fever, uncontrolled arrhythmias, uncompensated heart failure, acute pericarditis or myocarditis, recent thrombosis or thrombophlebitis, resting ST-segment deviation, uncontrolled diabetes, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
cardiopulmonary oxygen consumption | 12 weeks
  to observe the maximum exercise performance

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No